CLINICAL TRIAL: NCT01089998
Title: Open-label, Multicenter Study of the 18F-labeled PET/CT (Positron Emission Tomography / Computed Tomography) Tracer BAY86-9596 Following a Single Intravenous Administration of 200 or 300 MBq (Corresponding to ≤ 18 µg Mass Dose) for Evaluation of Radiation Dosimetry, Plasma Pharmacokinetics, Safety and Tolerability in Healthy Volunteers (200 MBq) as Well as Investigation of Safety, Tolerability and Diagnostic Performance in Patients (300 MBq) With Non-small Cell Lung Cancer, Breast Cancer, Head and Neck Cancer and in Patients With Inflammation.
Brief Title: PET/CT Imaging for Radiation Dosimetry, Plasma Pharmacokinetics, Safety and Tolerability in Healthy Volunteers and Safety, Tolerability and Diagnostic Performance of BAY86-9596 in Patients With Non-small Cell Lung Cancer, Breast Cancer, Head and Neck Cancer and Patients With Inflammations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14641; 2009-013098-16 (EudraCT Number)
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Diagnostic Imaging
Keywords: Neoplasm; PET/CT diagnosis; PET tracer; Inflammation
MeSH Terms: conditions — Neoplasms; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-9596
- Arm 2 (Experimental)
  Interventions: Drug: BAY86-9596
- Arm 3 (Experimental)
  Interventions: Drug: BAY86-9596
- Arm 4 (Experimental)
  Interventions: Drug: Fludeoxyglucose (18F)-IBA

INTERVENTIONS:
Drug: BAY86-9596 — Healthy volunteers, single intravenous bolus injection of 200 MBq BAY 86-9596 on day one of the treatment period, whole body PET/CT for determination of effective dose, kinetics of BAY 86-9596 in blood and urine
  Arms: Arm 1
Drug: BAY86-9596 — Cancer patients, single intravenous bolus injection of 300 MBq BAY 86-9596 on day one of the treatment period, PET/CT.
  Arms: Arm 2
Drug: BAY86-9596 — Inflammation patients, single intravenous bolus injection of 300 MBq BAY 86-9596 on day one of the treatment period, PET/CT.
  Arms: Arm 3
Drug: Fludeoxyglucose (18F)-IBA — Subgroup of cancer patients: radiation induced inflammation. Fluordeoxyglucose (18F)-FDG PET scan will be performed approx. 4 week after radiation and compared with tracer BAY86-9596 (acc. to Amendment 4 only in the Netherlands)
  Arms: Arm 4

SUMMARY:
Visual assessment of diagnostic PET/CT (positron emission tomography/computed tomography) images obtained after a single intravenous injection of BAY86-9596 in patients with cancer and inflammation

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers only

  * Males/females ≥ 50 years and ≤ 65 years of age
* Cancer patients and inflammation patients (inflammation patients in study part 2 = optional, in study part 3 mandatory)

  * Males/females ≥ 30 and ≤ 80 years of age
  * patients had an FDG PET/CT for detection, or staging, or restaging, or therapy response assessment that still showed tumor mass with high certainty, for

    1. NSCLC (non small cell lung cancer), or
    2. adenocarcinoma of the breast (female patients) or
    3. squamous cell cancer of head and neck and the cancer disease is histologically confirmed.
    4. Patients with confirmed/known inflammatory focus/foci after FDG-PET/CT imaging

Exclusion Criteria:

* Exclusion criteria for all healthy volunteers and patients:

  * any concomitant disease (for healthy volunteers) and for patients any concurrent severe and/or uncontrolled and/or unstable other medical disease (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of BAY86-9596, unstable and uncontrolled hypertension, chronic renal or hepatic disease, severe pulmonary disease) which could compromise participation in the study
  * For healthy volunteers and patients: known sensitivity to the study drug or components of the preparation.
  * tumor patients with known inflammatory disease, where images overlap inflammatory lesions with tumor lesions

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Visual assessment of lesions (tumor detection rate of BAY 86-9596 compared to FDG) | Day of study drug administration

SECONDARY OUTCOMES:
Quantitative analysis of BAY 86-9596 uptake into lesions (Standardized Uptake Values = SUVs) | Day of study drug administration
Vital signs (ECG, blood pressure, Heart rate, Body temperature) | At least 2 times within 8 days after treatment
Serum chemistry, Clotting status, Hematology | At least 2 times within 8 days after treatment
Adverse Event collection | At least 2 times within 8 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Groningen, Provincie Groningen, Netherlands
- Zurich, Canton of Zurich, Switzerland